CLINICAL TRIAL: NCT03850236
Title: Impact of the Neck Division Level During Pancreaticoduodenectomy on Postoperative Pancreatic Fistula?
Brief Title: Neck Division Level and Postoperative Pancreatic Fistula After Pancreaticoduodenectomy
Acronym: PaNECK
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0025
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Pancreatoduodenectomy
Keywords: pancreatic fistula; morbidity; risk factors; Benign or malign pathology
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Cytolyt Samples:
  Liquid conservation samples from patients who underwent endoscopic ultrasound with fine needle aspiration/biopsy for suspicious pancreatic mass at the CHU de Montpellier were conserved at +4°c.
  Cytolyt samples do not contain any cell or tissue from patient, this liquid is systematically trashed in current practice. No genetics analysis will be performed from these particular samples in the present study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief Summary:*

Aim of the study :

To evaluate if the neck division level significantly influences the postoperative pancreatic fistula rate of pancreatico-jejunal anastomosis after pancreatoduodenectomy.

Methods :

Patients who underwent oncologic or non-oncologic pancreatoduodenectomy between 01 January 2009 and 04 April 2018 will be included in this retrospective analysis. Two independent radiologists will measure the distance between the left side of the portal vein and the remnant pancreatic stump on post operative CT scan, blindly for postoperative course. This new variable will be integrated in a logistic regression model in addition to well known risk factors of POPF.

DETAILED DESCRIPTION:
The pancreatic neck is an anatomical area mainly vascularized by the arterial network derived from the gastroduodenal artery and branches of the superior mesenteric artery running in the pancreatic head.

The neck arterial blood supply is probably reduced after pancreatoduodenectomy due to the ligation of gastroduodenal artery and collaterals of superior mesenteric artery.

Postoperative pancreatic fistula (POPF) is the main complication after pancreatoduodenectomy. POPF has an estimated rate of 15 to 30%. So, this complication is frequent and could be lethal. Several studies have been driven to identify risks factors of POPF but there are no actual data on the impact of the neck division level and neck vascularization on POPF.

By considering the level of neck division is variable, the investigator hypothesize that a long remnant neck, is a risk factor of POPF after pancreatoduodenectomy with pancreatojejunal anastomosis.

The aim of the present study is to integrate this new variable in a logistic regression model in addition to well known risk factors of POPF.

ELIGIBILITY:
Inclusion criteria:

* Elective Pancreatoduodenectomy with pancreatojejunal anastomosis whatever the indication
* age > 18 y.o.

Exclusion criteria:

* past history of pancreatic surgery
* patient who reject the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring pancreatoduodenectomy for benign or malignant pathology.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
grade of fistula | 90 postoperative days
  fistula grade B / C pancreatico-jejunal anastomosis after cephalic duodeno-pancreatectomy

SECONDARY OUTCOMES:
Overall morbidity | 90 postoperative days
  Overall morbidity (according to Clavien Dindo Classification)

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

REFERENCES:
- [Derived] Bardol T, Delicque J, Hermida M, Herrero A, Guiu B, Fabre JM, Souche R. Neck transection level and postoperative pancreatic fistula after pancreaticoduodenectomy: A retrospective cohort study of 195 patients. Int J Surg. 2020 Oct;82:43-50. doi: 10.1016/j.ijsu.2020.08.001. Epub 2020 Aug 22. PMID 32841726